CLINICAL TRIAL: NCT00441285
Title: Antiparasitic Therapy for Neurocysticercosis: Phase II/III Study on Safety and Efficacy of Combined Treatment With Praziquantel and Albendazole
Brief Title: Neurocysticercosis: Combined Treatment With Praziquantel (PZQ) and Albendazole (ABZ)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01NS054805 (NIH); R01NS054805 (NIH)
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-05

CONDITIONS: Neurocysticercosis; Epilepsy
Keywords: neurocysticercosis; NCC; praziquantel; PZQ; albendazole; ABZ; parasite; pig tapeworm; Taenia solium; epilepsy; late-onset epilepsy; acquired epilepsy
MeSH Terms: conditions — Neurocysticercosis; Epilepsy; Taeniasis | interventions — Praziquantel; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I. ABZ + ABZ Placebo + PZQ (Active Comparator): Albendazole 15 mg / kg / d (until 800 mg / d) + Placebo of Albendazole ( 7.5 mg / Kg / d )+ Praziquantel 50 mg / kg / d (until 3600 mg / d)
  Interventions: Drug: Praziquantel; Drug: Albendazole; Drug: ABZ Placebo
- II.- ABZ + ABZ Placebo + PZQ Placebo (Active Comparator): Albendazole 15 mg / kg / d ( until 800 mg / d ) + Placebo of Albendazole ( 7.5 mg / Kg / d ) + Placebo of Praziquantel ( 50 mg / kg / d )
  Interventions: Drug: Albendazole; Drug: ABZ Placebo; Drug: PZQ Placebo
- III .- Albendazole + PZQ Placebo (Active Comparator): Albendazole 22.5 mg / kg / d (until 1200 mg / d) + Placebo of Praziquantel ( 50 mg / kg / d )
  This arm was not used in the first substudy ( initial part and guide to the design of the parent study ) however it will be used henceforward.
  Interventions: Drug: Albendazole; Drug: PZQ Placebo

INTERVENTIONS:
Drug: Praziquantel — - Praziquantel 50 mg / kg / d (up to 3600 mg / d ) for 10 days.
  Other Names: PZQ
  Arms: I. ABZ + ABZ Placebo + PZQ
Drug: Albendazole — * Albendazole 15 mg / kg / d ( up to 800 mg /d ) in Arm I for 10 days.
  * Albendazole at an increased dose, 22.5 mg / kg / d (up to 1200 mg / d ), in Arm II for 10 days.
  Other Names: ABZ
Drug: ABZ Placebo — - Placebo (of Albendazole ) 7.5 mg / kg / d in Arm I and II for 10 days.
  Other Names: Placebo of Albendazole
  Arms: I. ABZ + ABZ Placebo + PZQ; II.- ABZ + ABZ Placebo + PZQ Placebo
Drug: PZQ Placebo — - Placebo (of Praziquantel) 50 mg / kg / d in Arm II and III for 10 days.
  Other Names: Placebo of PZQ
  Arms: II.- ABZ + ABZ Placebo + PZQ Placebo; III .- Albendazole + PZQ Placebo

SUMMARY:
The purpose of this study is to determine if combination drug therapy of praziquantel and albendazole is safe and effective to cure neurocysticercosis.

DETAILED DESCRIPTION:
Neurocysticercosis is the single major cause of acquired or late-onset epilepsy in the world, and a common diagnosis in immigrant populations in the United States and other industrialized countries. An estimated 50 million humans are affected by Neurocysticercosis. The disease occurs when a parasite called Taenia solium, or the pig tapeworm, infects the brain, forming cysts. Neurocysticercosis is generally treated with 1 of 2 drugs, praziquantel or albendazole. However, current treatment with either of these drugs alone is not totally effective.

The goal of this trial is to determine if combination drug therapy of praziquantel and albendazole is safe and more effective to cure Neurocysticercosis than either drug administered alone. This trial will consist of two sub-studies and a parent study.

In the first substudy which was performed and completed as the initial part and guide to the design of the parent study, a series of 32 patients with viable cystic intraparenchymal Neurocysticercosis were treated with either albendazole ( 15 mg / kg /d ) + praziquantel ( 50 mg / kg/ d ) or albendazole+Placebo in a double blind randomized study. Half of patients in each group had their seizure disorder treated with phenytoin and the other half with carbamazepine (not assigned by the study). The study was designed and powered for pharmacokinetic evaluation and exploratory safety so comparative cysticidal efficacy has not yet been analyzed. There were no safety concerns. Pharmacokinetics of ABZ and PZQ were obtained and described.

In the parent study, a total of 240 participants ( including the 32 participants from the first substudy ) will be randomly chosen to receive albendazole + praziquantel, albendazole + placebo or albendazole at an increased dose + placebo for 10 days. These groups will also receive other standard medications to manage the disease including appropriate anti-epileptic drug therapy. Participants will stay in the hospital for at least 2 weeks after treatment begins, which includes 5 days after the end of anti-parasitic treatment. After discharge from the hospital, follow-up visits will be on days 21 and 30 after treatment begins, then monthly until day 90, and finally every 3 months until completing 18 months. Brain images will be taken at 6 and 12 months after treatment begins. For participants, duration of the trial is 1 year and a half.

ELIGIBILITY:
For parent study:

Inclusion Criteria:

* Male or female individuals between 16 to 65 years of age, with a diagnosis of Neurocysticercosis and 20 or less viable cysts.
* Patients with a diagnosis of epilepsy secondary to Neurocysticercosis and a history of one or more spontaneous seizures within the previous year but not longer than 10 years.
* Willingness to complete a minimum of two weeks of hospitalization.
* If female of child bearing potential, negative urine pregnancy testing and willingness to use an adequate method of contraception while on study medications and for at least 3 months following Albendazole therapy.
* Normal laboratory values for hematocrit, platelets, white blood cells and glucose and normal or decreased values for Alanine transaminase, Aspartate transaminase and creatinine.
* Negative PPD measurement and if positive ( > 9mm induration in the absence of other findings or immunosuppression ) , negative smears for TB.
* Negative fecal exam for Taenia eggs or Strongyloides larvae.

Exclusion Criteria:

* Primary generalized seizures ( e.g., not caused by Neurocysticercosis )
* A history of generalized epileptic status .
* A type of Neurocysticercosis which can expose the patient to increased risk during the study.
* Patients with persistent or progressive symptomatic intracranial hypertension or intracranial hypertension.
* Previous therapy with Albendazole or Praziquantel in the previous year.
* Pulmonary tuberculosis, or symptoms compatible with tuberculosis not otherwise explained.
* Active hepatitis
* Systemic disease that may affect short term prognosis.
* Patients in unstable condition ( consistently abnormal vital signs: body temperature, heart rate, respiratory rate, and blood pressure )
* Pregnancy during antiparasitic treatment
* History of hypersensitivity to Albendazole or Praziquantel
* Concurrent treatment with Cimetidine or Theophylline
* Chronic alcohol or drug abuse
* Unwilling or unable to provide a Computed tomography initially or an Magnetic resonance imaging at 6 months ( as patients with ferromagnetic implants ) , Computed tomography at the end of therapy.
* Unwillingness of subject or legal representative to give written informed consent.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector H. Garcia, MD, Principal Investigator — Universidad Peruana Cayetano Heredia; E. Javier Pretell, MD, Principal Investigator — Hospital Alberto; Javier A. Bustos, MD, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (5):
- Peru (5):
  - Hospital Nacional Edgardo Rebagliati, Lima, Lima Province
  - Hospital Nacional Cayetano Heredia, Lima, Lima Province
  - Hospital Nacional Guillermo Almenara, Lima, Lima Province
  - Instituto Nacional de Ciencias Neurologicas, Lima
  - Universidad Peruana Cayetano Heredia, Lima

REFERENCES:
- [Result] Garcia HH, Lescano AG, Lanchote VL, Pretell EJ, Gonzales I, Bustos JA, Takayanagui OM, Bonato PS, Horton J, Saavedra H, Gonzalez AE, Gilman RH; Cysticercosis Working Group in Peru. Pharmacokinetics of combined treatment with praziquantel and albendazole in neurocysticercosis. Br J Clin Pharmacol. 2011 Jul;72(1):77-84. doi: 10.1111/j.1365-2125.2011.03945.x. PMID 21332573
- [Result] Garcia HH, Gonzales I, Lescano AG, Bustos JA, Zimic M, Escalante D, Saavedra H, Gavidia M, Rodriguez L, Najar E, Umeres H, Pretell EJ; Cysticercosis Working Group in Peru. Efficacy of combined antiparasitic therapy with praziquantel and albendazole for neurocysticercosis: a double-blind, randomised controlled trial. Lancet Infect Dis. 2014 Aug;14(8):687-695. doi: 10.1016/S1473-3099(14)70779-0. Epub 2014 Jul 3. PMID 24999157
- [Derived] Garcia HH, Lescano AG, Gonzales I, Bustos JA, Pretell EJ, Horton J, Saavedra H, Gonzalez AE, Gilman RH; Cysticercosis Working Group in Peru. Cysticidal Efficacy of Combined Treatment With Praziquantel and Albendazole for Parenchymal Brain Cysticercosis. Clin Infect Dis. 2016 Jun 1;62(11):1375-9. doi: 10.1093/cid/ciw134. Epub 2016 Mar 16. PMID 26984901

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol (2 groups, n=180) was modified by the DSMB to add a pharmacokinetics / safety substudy (two groups, n=32). After the substudy results were available, we were approved to proceed with a modified study design (3 groups, n=240). This second study was terminated after enroling patient 124 because of early efficacy (total n= 132+24, 156)
Groups:
- PK Substudy ABZ+PZQ: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * Praziquantel was given at 50 mg / kg / d , divided in two daily doses, morning and evening.It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g / d , for 9 1/2 days.
- PK Substudy ABZ+Placebo: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * Praziquantel placebo was given in two daily doses, morning and evening,for 9 1/2 days.
- Phase III Trial - ABZ+PZQ: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * Placebo of ABZ was added to mask the dose of ABZ (see Increased ABZ arm)
  * Praziquantel was given at 50 mg / kg / d , divided in two daily doses, morning and evening.It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g / d , for 9 1/2 days.
- Phase III Trial - Increased ABZ: * Albendazole was given at 22.5 mg / kg / d , divided in two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum of 1200 mg / d, for 10 days.
  * Praziquantel was given at 50 mg / kg / d , divided in two daily doses, morning and evening. It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g / d , for 9 1/2 days.
- Phase III Trial - Standard ABZ: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * Placebo of ABZ was added to mask the dose of ABZ (see Increased ABZ arm)
  * Placebo of Praziquantel was given at 50 mg / kg / d , divided in two daily doses, morning and evening.It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g / d , for 9 1/2 days.
Period: Overall Study
Arm/Group | PK Substudy ABZ+PZQ | PK Substudy ABZ+Placebo | Phase III Trial - ABZ+PZQ | Phase III Trial - Increased ABZ | Phase III Trial - Standard ABZ
Started | 16 | 16 | 41 | 40 | 43
Completed | 16 | 16 | 41 | 40 | 43
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The population involves 32 patients in the Phase II substudy and 124 patients in the Phase III main study
Groups:
- Albendazole + Praziquantel: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * Praziquantel was given at 50 mg / kg / d , divided in two daily doses, morning and evening.It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g / d , for 9 1/2 days.
- Albendazole + Placebo: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * Praziquantel placebo was given in two daily doses, morning and evening,for 9 1/2 days.
- Phase III Trial ABZ+PZQ: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * A placebo of ABZ was added to complete to the doses in the Increased ABZ arm
  * Praziquantel was given at 50 mg / kg / d , divided in two daily doses, morning and evening.It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g / d , for 10 days.
- Phase III Trial Increased ABZ: * Albendazole was given at 22.5 mg / kg / d , divided in two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum of 1200 mg / d , for 10 days.
  * Praziquantel placebo was given in two daily doses, morning and evening,for 10 days.
- Phase III Trial Standard ABZ: * Albendazole was given at 15 mg / kg / d , divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg / d , for 10 days.
  * A placebo of ABZ was added to complete the doses to the dosage in the Increased ABZ arm
  * Praziquantel placebo was given in two daily doses, morning and evening,for 10 days.
- Total: Total of all reporting groups
Arm/Group | Albendazole + Praziquantel | Albendazole + Placebo | Phase III Trial ABZ+PZQ | Phase III Trial Increased ABZ | Phase III Trial Standard ABZ | Total
Number analyzed (Participants) | 16 | 16 | 41 | 40 | 43 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 0 | 2 | 2 | 8
  Between 18 and 65 years | 14 | 14 | 39 | 38 | 41 | 146
  >=65 years | 0 | 0 | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (9.7) | 27.5 (11) | 34 (14) | 34 (12) | 35 (13) | 28 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 15 | 19 | 14 | 59
  Male | 11 | 10 | 26 | 21 | 29 | 97
Region of Enrollment [Number; unit: participants]
  Peru | 16 | 16 | 41 | 40 | 43 | 156

OUTCOME MEASURES:

1. Primary Outcome: PK Substudy - Area Under the Curve of Albendazole in Treatment in Day 1
Description: - To evaluate kinetic disposition of Albendazole we calculated the Area under the curve of the active metabolite of Albendazole (Albendazole Sulphoxide) with Praziquantel or Placebo (of Praziquantel).
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 10 and 12 hours post dose on Treatment day 1
Measure: Mean (95% Confidence Interval); unit: ng*h/mL
Arm/Group | Albendazole + Praziquantel | Albendazole + Placebo
Number analyzed (Participants) | 16 | 16
ng*h/mL | 1412.2 (58124.7) [1115.5 to 1709] | 1111 (32257.1) [931.1 to 1290.8]

2. Primary Outcome: PK Substudy - Area Under the Curve of Albendazole in Treatment Days 10 and 11
Description: as for outcome 1
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 8, 10, 12, 24 and 36 hours post dose on Treatment days 10-11
Measure: Mean (95% Confidence Interval); unit: ng*h/ml
Arm/Group | Albendazole + Praziquantel | Albendazole + Placebo
Number analyzed (Participants) | 16 | 16
ng*h/ml | 4925.3 [3548.6 to 6302] | 2969.6 [2543.8 to 3395.4]

3. Secondary Outcome: PK Substudy - Area Under the Curve of Praziquantel by Antiepileptic Drug in Treatment Day 1
Description: - To evaluate the kinetic disposition of Praziquantel by antiepileptic drug after the last praziquantel dose, we calculated the Area Under the Curve of Praziquantel with Carbamazepine or Phenytoin
Time Frame: 0, 0.5, 1, 1.5, 2, 3, 4, 8, 10 and 12 hours post dose in treatment day 1
Population: Carbamazepine and Phenytoin were not assigned by the study.
Measure: Mean (Standard Deviation); unit: ng*h / mL
Groups:
- Albendazole + Praziquantel: * Albendazole was given at 15 mg/kg/day, divided two daily doses, morning and evening. It is supplied in 200 mg tablets, so the dose was rounded up to the next 100 mg level, up to a maximum 800 mg/day, for 10 days.
  * Praziquantel was given at 50 mg/kg/day, divided in two daily doses, morning and evening.It is supplied in 600 mg tablets divided in four, so the dose was rounded up to the next 100 mg level, up to a maximum 3.6 g/day,for 9 1/2 days.
Arm/Group | Albendazole + Praziquantel
Number analyzed (Participants) | 16
ng*h / mL
  Carbamazepine (n=8) | 548.3 (320.9)
  Phenytoin (n=8) | 923.7 (424.7)

4. Secondary Outcome: PK Substudy - Area Under the Curve of Praziquantel by Antiepileptic Drug in Treatment Days 10 and 11
Description: as for outcome 3
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 8, 10, 12, 24 and 36 hours post dose on treatment days 10-11
Measure: Mean (95% Confidence Interval); unit: ng*h/ml
Groups:
- Carbamazepine: Area Under the Curve of Praziquantel in Patients Receiving Carbamazepine
- Phenytoin: Area Under the Curve of Praziquantel in Patients Receiving Phenytoin
Arm/Group | Carbamazepine | Phenytoin
Number analyzed (Participants) | 8 | 8
ng*h/ml | 240.2 [151.7 to 328.7] | 550.1 [83.3 to 1183.4]

5. Primary Outcome: PK Substudy - Maximum Concentration of Albendazole
Description: Highest serum level of Albendazole measured from all level assessments in the curve.
Time Frame: Treatment day 1 and Treatment days 10-11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Albendazole + Praziquantel | Albendazole + Placebo
Number analyzed (Participants) | 16 | 16
ng/mL | 1293.9 (3471.6) | 2232.8 (6500.7)

6. Secondary Outcome: PK Substudy - Safety of Combined Albendazole Plus Praziquantel Therapy
Description: - Describe if some Serious Adverse Event was associated to combined Albendazole plus Praziquantel therapy.
Time Frame: 90 days post tx
Measure: Number; unit: Events
Arm/Group | Albendazole + Praziquantel | Albendazole + Placebo
Number analyzed (Participants) | 16 | 16
Events | 0 | 0

7. Secondary Outcome: Phase III Trial - Proportion of Cysts Which Resolved
Description: Proportion of Viable Brain Parasites which Are not Alive Anymore at 6 Months MRI
Time Frame: Day 180
Population: Final population numbers for this analysis not yet defined
Groups:
- Phase III Trial - ABZ+PZQ: Main Trial, Arm receiving standard ABZ doses plus active PZQ
- Phase III Trial - Increased ABZ: Main Trial, Arm receiving increased ABZ doses, no PZQ
- Phase III Trial - Standard ABZ: Main Trial, Arm receiving standard ABZ doses, no PZQ
Arm/Group | Phase III Trial - ABZ+PZQ | Phase III Trial - Increased ABZ | Phase III Trial - Standard ABZ
Number analyzed (Participants) | 0 | 0 | 0

8. Primary Outcome: Phase III Trial - Proportion of Patients Without Remaining Live Cysts
Description: Proportion of patients whose 6 month MR does not show viable parasites anymore
Time Frame: Day 180
Population: Some patients did not reach the analysis time point.
Measure: Number; unit: participants
Arm/Group | Phase III Trial - ABZ+PZQ | Phase III Trial - Increased ABZ | Phase III Trial - Standard ABZ
Number analyzed (Participants) | 39 | 38 | 42
participants | 25 | 19 | 15

9. Secondary Outcome: Phase III Trial - Seizure Frequency
Description: Seizure frequency by treatment group
Time Frame: Day 1 - 540
Population: Final population numbers for this analysis not yet defined
Arm/Group | Phase III Trial - ABZ+PZQ | Phase III Trial - Increased ABZ | Phase III Trial - Standard ABZ
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Number of Serious Adverse Events along the entire follow up (Days 1 - 540)
Description: Adverse events by treatment arm in Phase III arms are not yet available because of the blinded nature of the trial
Arm/Group | Albendazole + Praziquantel | Albendazole + Placebo
Serious Adverse Events (participants affected / at risk) | 2/16 | 2/16
Other Adverse Events (participants affected / at risk) | 15/16 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole + Praziquantel (N=16) | Albendazole + Placebo (N=16)
Prolonged hospitalization (Nervous system disorders) | 2 (2) | 2 (2) — The Prolonged hospitalization was associated with the disease itself, not because of antiparasitic treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole + Praziquantel (N=16) | Albendazole + Placebo (N=16)
Headache (Nervous system disorders) | 4 (6) | 5 (9)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Decreased indirect bilirubin (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased neutrophilos (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Decreased Red blood cells (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Decreased White blood cells (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Hypoesthesia (Nervous system disorders) | 0 (0) | 3 (4)
Increased ALT (Gastrointestinal disorders) | 8 (9) | 10 (17)
Increased AST (Gastrointestinal disorders) | 3 (3) | 7 (9)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes